CLINICAL TRIAL: NCT01048892
Title: A Phase 1 Dose Escalation Study of Seneca Valley Virus (NTX-010), A Replication-Competent Picornavirus, in Relapsed/Refractory Pediatric Patients With Neuroblastoma, Rhabdomyosarcoma, or Rare Tumors With Neuroendocrine Features
Brief Title: Seneca Valley Virus-001 and Cyclophosphamide in Treating Young Patients With Relapsed or Refractory Neuroblastoma, Rhabdomyosarcoma, or Rare Tumors With Neuroendocrine Features
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADVL0911; COG-ADVL0911; CDR0000663520 (Other: Clinical Trials.gov)
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Adrenocortical Carcinoma; Gastrointestinal Carcinoid Tumor; Kidney Cancer; Neuroblastoma; Retinoblastoma; Sarcoma
Keywords: recurrent neuroblastoma; previously treated childhood rhabdomyosarcoma; recurrent childhood rhabdomyosarcoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent retinoblastoma; recurrent adrenocortical carcinoma; recurrent gastrointestinal carcinoid tumor
MeSH Terms: conditions — Adrenocortical Carcinoma; Kidney Neoplasms; Neuroblastoma; Retinoblastoma; Sarcoma; Wilms Tumor | interventions — Cyclophosphamide

ARMS (1):
- Treatment (NTX-010) (Experimental)
  Interventions: Biological: Seneca Valley virus-001; Drug: cyclophosphamide; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: Seneca Valley virus-001
Drug: cyclophosphamide
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Seneca Valley virus-001 may be able to kill certain kinds of tumor cells without damaging normal cells. Adding low dose cyclophosphamide (in part B of study) may help to kill even more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of Seneca Valley virus-001 in treating young patients with relapsed or refractory neuroblastoma, rhabdomyosarcoma, or rare tumors with neuroendocrine features.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the maximum-tolerated dose and/or recommended phase II dose of Seneca Valley virus-001 (NTX-010) when administered as a single infusion to pediatric patients with relapsed or refractory neuroblastoma, rhabdomyosarcoma, or rare tumors with neuroendocrine features (Wilms tumor, retinoblastoma, adrenocortical carcinoma, or carcinoid tumors). (Part A [completed])
* To confirm that there is viral replication in these patients following NTX-010 administration. (Part A [completed])
* To define and describe the toxicities of NTX-010 when administered on this schedule. (Part A [completed])
* To determine whether the number of regulatory T cells (as measured by flow cytometry) can effectively be reduced following administration of NTX-010 plus low-dose metronomic and intravenous cyclophosphamide. (Part B)
* To characterize the pharmacokinetics (time course of viral clearance) following NTX-010 administration in these patients.

Secondary

* To preliminarily define the antitumor activity of NTX-010 within the confines of a phase I study. (Part A [completed])
* To evaluate the development of neutralizing antibodies to NTX-010 following IV administration of NTX-010. (Part A [completed])
* To evaluate development of neutralizing antibodies to NTX-010 following the combination of NTX-010 and cyclophosphamide. (Part B)
* To investigate the presence and permissivity of occult circulating tumor cells prior to and after the initial intravenous administration of NTX-010.

OUTLINE: This is a multicenter study.

Part A (completed): Patients receive Seneca Valley virus-001 (NTX-010) IV over 1 hour on day 1.

Part B: Patients receive cyclophosphamide IV orally (PO) on days 1-14 and NTX-010 IV over 1 hour on day 8. In the absence of disease progression or unacceptable toxicity, patients then receive cyclophosphamide orally (PO) on days 22-35, plus cyclophosphamide IV over 1 hour and NTX-010 IV over 1 hour on day 29.

Tumor tissue samples are collected at baseline for biomarker studies. Blood and stool samples are collected periodically for neutralizing antibody and viral clearance studies. Additional blood samples may also be collected for the presence and permissivity of occult tumor cells.

After completion of study treatment, patients are followed up periodically for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of 1 of the following:

  * Neuroblastoma
  * Rhabdomyosarcoma
  * Wilms tumor
  * Retinoblastoma
  * Adrenocortical carcinoma
  * Carcinoid tumor
* Relapsed or refractory disease
* Measurable or evaluable disease
* No known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* No known pulmonary tumors or metastases > 5 cm, as evaluated by chest CT scan
* No clinically significant pulmonary and/or pericardial effusions (≥ grade 3), as evaluated by ECHO
* No primary CNS tumors or known metastatic CNS disease involvement

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 50-100% (for patients > 16 years of age)
* Lansky PS 50-100% (for patients ≤ 16 years of age)
* Peripheral ANC ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent, defined as no platelet transfusions within a 7-day period before study enrollment)
* Hemoglobin ≥ 8.0 g/dL (RBC transfusions allowed)
* Creatine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * ≤ 0.8 mg/dL (for patients 3 to 5 years of age)
  * ≤ 1.0 mg/dL (for patients 6 to 9 years of age)
  * ≤ 1.2 mg/dL (for patients 10 to 12 years of age)
  * ≤ 1.4 mg/dL (for female patients ≥ 13 years of age)
  * ≤ 1.5 mg/dL (for male patients 13 to 15 years of age)
  * ≤ 1.7 mg/dL (for male patients ≥ 16 years of age)
* Bilirubin (sum of conjugated and unconjugated) ≤ 1.5 times upper limit of normal (ULN)
* SGPT ≤ 110 U/L (for the purpose of this study, the ULN for SGPT is 45 U/L)
* Serum albumin ≥ 2 g/dL
* Oxygen saturation > 92% on room air
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to comply with the safety monitoring requirements of the study, in the opinion of the investigator
* Completely toilet trained
* No chronic diarrhea or urinary incontinence during the day or night, , and no in-dwellling urinary catheters
* No uncontrolled infection
* No known pregnant member of the household

PRIOR CONCURRENT THERAPY:

* Fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy
* At least 6 months since prior total-body irradiation (TBI), craniospinal radiotherapy, or radiotherapy to ≥ 50% of the pelvis
* At least 3 months since prior stem cell transplantation or rescue (without TBI)

  * No evidence of active graft-vs-host disease
* At least 6 weeks since other prior substantial bone marrow radiotherapy or treatment with therapeutic doses of MIBG
* More than 3 weeks since prior myelosuppressive chemotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* More than 7 days since prior growth factor(s) that support platelet or white blood cell number or function
* At least 7 days since prior biologic agents
* At least 3 half-lives since prior monoclonal antibodies
* More than 7 days since prior viral immunizations, including influenza
* At least 42 days since the completion of any type of immunotherapy, e.g., tumor vaccines
* No other viral immunizations after enrolling on study until 28 days after their last planned Seneca Valley virus-001 infusion or until documented viral clearance, whichever is longest
* Concurrent corticosteroids allowed provided the patient has been on a stable or decreasing dose for the past 7 days
* No other concurrent investigational drugs
* No other concurrent anticancer agents (e.g., chemotherapy, radiotherapy, immunotherapy, or biologic therapy)
* Prior treatment with Seneca Valley virus-001 is not allowed

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 12 months post-documented viral clearance
Recommended phase II dose of Seneca Valley virus-001 (NTX-010) | 56 days

SECONDARY OUTCOMES:
Tumor response | Up to 12 months post documented viral clearance
Viral titers in blood and stool | Up to 56 days post treatment
Development of antibodies to NTX-010 | Up to 4 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Burke, MD, Study Chair — Masonic Cancer Center, University of Minnesota
Locations (18):
- United States (18):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Riley's Children Cancer Center at Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin